CLINICAL TRIAL: NCT00008190
Title: High Dose Chemotherapy And Autologous Peripheral Blood Stem Cell Rescue For High Risk Acute Leukemia
Brief Title: Combination Chemotherapy Followed by Peripheral Stem Cell Transplantation and Interleukin-2 in Treating Patients With Acute Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068386; CPMC-IRB-8872; CPMC-CAMP-27; NCI-G00-1889
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2004-04

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — aldesleukin; Filgrastim; Busulfan; Cyclophosphamide; Etoposide; Melphalan; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: aldesleukin
Biological: filgrastim
Drug: busulfan
Drug: cyclophosphamide
Drug: etoposide
Drug: melphalan
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Interleukin-2 may stimulate a person's white blood cells to kill leukemia cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by peripheral stem cell transplantation and interleukin-2 in treating patients who have acute leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of busulfan, cyclophosphamide, and etoposide followed by autologous peripheral blood stem cell transplantation and interleukin-2 in patients with high-risk acute leukemia.
* Determine the efficacy of immunomodulatory therapies in terms of relapse-free survival of these patients treated with this regimen.
* Determine the hematopoietic reconstitution, relapse, and survival of these patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Following a course of mobilization chemotherapy, patients receive priming therapy comprising filgrastim (G-CSF) and interleukin-2 through the completion of leukapheresis. Patients then receive oral busulfan 4 times daily on days -8 through -5, cyclophosphamide IV continuously on days -4 and -3, and etoposide IV over 2 hours on day -4. For patients unable to receive cyclophosphamide and etoposide, melphalan IV is administered instead on days -3 and -2. Autologous peripheral blood stem cells (PBSC) are reinfused on day 0.

Patients then receive G-CSF daily beginning on day 0 and continuing until blood counts recover followed by interleukin-2 subcutaneously daily beginning at the completion of G-CSF therapy and continuing for 6 months.

Patients are followed weekly for 1 month and then monthly thereafter.

PROJECTED ACCRUAL: A total of 19-25 patients will be accrued for this study within 3-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed acute leukemia

  * High-risk due to any of the following:

    * Cytogenetic abnormalities involving 5q, 7q, 8q, 11q23, or t(9;22)
    * WBC greater than 100,000/mm3
    * Prior myelodysplastic syndrome
    * Complete remission (CR) lasting less than 12 months
  * No favorable cytogenetic parameters (e.g., t(15;17), inv16, or t(8;21))
* CR following standard anti-leukemic therapy confirmed by bone marrow evaluation

  * Second and third CR allowed
* Ineligible for higher priority national or institutional study or allogeneic peripheral blood stem cell transplantation

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin less than 1.5 times normal
* SGOT or SGPT less than 1.5 times normal

Renal:

* Creatinine less than 1.5 times normal

Cardiovascular:

* LVEF at least 45% if receiving cyclophosphamide
* Normal electrocardiogram OR
* Approval by cardiologist

Pulmonary:

* DLCO less than 60% predicted OR
* Approval by pulmonologist

Other:

* Not pregnant or nursing
* No concurrent illness that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-03; Primary Completion 2005-11 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Hesdorffer, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States